CLINICAL TRIAL: NCT00861822
Title: Advance Targeted Transfusion in Anemic Cardiac Surgical Patients for Kidney Protection: A Proof of Concept Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-1083-B
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Injury
Keywords: Anemia; Cardiac surgery; RBC transfusion; Acute Kidney Injury; Cardiac surgery with cardiopulmonary bypass
MeSH Terms: conditions — Anemia; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RBC (Active Comparator): Advance RBC transfusion' (ART) group
  Interventions: Other: Advanced red blood cell transfusion
- Standard Care (Other): Standard-of-care RBC transfusion (SRT) group
  Interventions: Other: Advanced red blood cell transfusion

INTERVENTIONS:
Other: Advanced red blood cell transfusion — Sixty anemic (Hg 100-120 g/L) adult patients undergoing cardiac surgery with CPB will be randomized to the 'advance RBC transfusion' (ART) group or the standard-of-care RBC transfusion' (SRT) group (1:1 ratio).
  In the ART group, subjects will receive 1-2 units of stored RBCs 1-2 days before surgery to reach a target Hb of 130-140 g/L. Each unit of blood will be transfused over 2 hours under medical supervision, with appropriate monitoring and management of fluid status to ensure patients are not over-hydrate

SUMMARY:
One of the major complications of heart surgery is kidney injury, which occurs in up to 30% of patients and is associated with poor outcomes including death. We have found that patients whose hemoglobin concentration before surgery is lower than normal (i.e., are anemic) are at particularly high risk for this complication, likely because their hemoglobin concentration drops to very low levels during surgery, which reduces delivery of oxygen to the kidneys, increases blood loss, and necessitates blood transfusions. We and others have shown that these events are individually harmful to the kidneys, and can lead to kidney injury. We believe that we can prevent these events from occurring, and as a result reduce the risk of kidney injury, if we transfuse anemic patients at least 1 day before surgery rather than during surgery.

In anemic patients undergoing cardiac surgery, prophylactic transfusion of red blood cells (RBCs) before surgery will reduce the risk of acute kidney injury (AKI) after surgery by mitigating three inter-related risk factors for AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-emergent aortocoronary bypass (ACB) surgery, or valve surgery, combined ACB and valve, or aortic root repair requiring CPB with a preoperative Hb concentration between 100 and 120 g/L.

Exclusion Criteria:

* Any conditions that may limit the ability of patients to tolerate the intervention:
* Severe aortic or mitral valve stenosis
* History of congestive heart failure within 30 days of surgery or severe ventricular dysfunction (ejection fraction < 30%)
* Severe (> 60%) left main coronary artery stenosis or unstable angina within 30 days of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effects on perioperative (within 72 hours of termination of CPB) anemia will be measured by: incidence of profound perioperative anemia (Hb < 70 g/L) and by nadir perioperative Hb concentration. | preoperatively, intraoperatively, postoperatively, daily until discharge

SECONDARY OUTCOMES:
(Primary)Effects on periop RBC transfusion rates measured by: incidence and amount of periop RBC transfusions. Effects on periop coagulation measured by: incidence and amount of coagulation product transfusions and incidence of surgical re-exploration. | preoperatively, intraoperatively, postoperatively, daily until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — Toronto General Hospital, Toronto, Ontario,Canada
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada